CLINICAL TRIAL: NCT06172374
Title: DNAI1 Primary Ciliary Dyskinesia: Genetic Testing, Patient Finding and Increasing Disease Awareness Program
Brief Title: A Study Providing Genetic Testing to Find Those Who May Have Primary Ciliary Dyskinesia for Potential Clinical Trials
Status: Active, not recruiting | Type: Observational
Sponsor: ReCode Therapeutics (Industry)
Collaborators: Sano Genetics (Industry); Reverba (Unknown)
Responsible Party: Sponsor
Other Study IDs: thinkPCD
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PCD Individuals confirmed positive for DNAI1
  Interventions: Genetic: Sano Genetics Testing Kit
- PCD Individuals confirmed positive for other genotypes of interest
  Interventions: Genetic: Sano Genetics Testing Kit
- Individuals negative for a gene causing PCD
  Interventions: Genetic: Sano Genetics Testing Kit

INTERVENTIONS:
Genetic: Sano Genetics Testing Kit — Genetic testing spit collection tubes for DNA testing

SUMMARY:
Primary purpose is to identify individuals who have PCD due to a genetic mutation within the DNAI1 and other genes of interest to help refer participants to future clinical studies for this rare disease.

DETAILED DESCRIPTION:
The aim of this study is to identify individuals with Primary ciliary dyskinesia (PCD) through a screening questionnaire that enriches for likely pathogenic gene mutations in DNAI1 and other genes of interest associated with PCD. Identified individuals will be referred to relevant upcoming clinical trials. This study will also obtain information on the proportion of individuals with PCD who have mutations in DNAI1, and other PCD genes of interest. Additional goals include increasing the awareness of patients and healthcare providers (HCPs) of the importance of genetic testing in PCD, and engaging their interest in future clinical studies.

PCD is a genetically heterogenous disease characterized by impaired ciliary movement in the lungs, paranasal sinuses, reproductive system, and Eustachian tubes. PCD can result in a range of clinical presentations, including pulmonary disease and respiratory tract infections, chronic sinus infections, and recurrent ear infections, among others. The estimated incidence of PCD is one in 10,000 people. Mutations in over 40 genes have been shown to cause PCD, with commonly implicated genes being DNAH5, DNAI1, and DNAH11.

There is currently a lack of effective diagnostic tools for PCD; an estimated 46,000 people with PCD remain undiagnosed in the United States. Genetic testing represents a potential method to diagnose PCD.

Individuals with a confirmed PCD diagnosis, or those strongly suspected to have PCD by HCPs, will complete an online informed consent form and a questionnaire to identify pathogenic mutations. Following consent, individuals will be sent no-cost genetic testing kits and guidance on collecting saliva samples. The saliva samples will be assessed by whole exome sequencing for a number of the genes implicated in PCD, including DNAI1. Individuals with identified DNAI1 mutations will be referred to the ReCode Therapeutics, Inc.'s RCT1100 Virtual Waiting Room and retained for potential future clinical trials through a continuing engagement scheme. Individuals with other PCD-causing mutations will also be retained for potential future clinical trials. Counselling will be available to all individuals in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years old.
2. Participant must have a prior diagnosis of PCD or be deemed eligible upon completion of the PCD-enrichment screening questionnaire.
3. Participant must be under the care of an HCP for their PCD or symptoms potentially related to PCD.
4. Participant must be able to read, write, and understand English, and reside in a country where the shipment of biological samples is allowed.
5. Participant must be willing to be tested for genes involved in PCD.
6. Participant must be willing to be notified of eligibility for clinical studies (if appropriate)

Exclusion Criteria:

In ability to meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with pathogenic mutation of genes known to cause PCD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of PCD individuals with DNAI1 mutation identified through genetic testing | 2 years
  Number of individuals with DNAI1 will be measured by tracking amount of completed questionnaires eligible for genetic testing resulting with DNAI1 gene mutation

SECONDARY OUTCOMES:
Proportion of PCD individuals with DNAI1 mutations and number of patients with mutations in other PCD genes of interest | 2 years
  Number of identified genotypes, including DNAI1, will be confirmed by analyzed saliva samples submitted from eligible individuals
Number of Health Care Provider (HCP) and their referred individuals eligible for genetic testing for PCD | 2 years
  Number of HCP and potential patients will be measured by number of questionnaires confirming eligibility for genetic testing for PCD

CONTACTS AND LOCATIONS:
Overall Officials: John G. Matthews, MBBS, MRCP, PhD, Study Chair — ReCode Therapeutics, Inc.
Locations (1):
- ReCode Therapeutics, Inc., Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No